CLINICAL TRIAL: NCT04396977
Title: Inter-arm and Inter-period Reproducability of the Dermal Blood Flow Response After a Histamine Skin Prick.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CCP18-3305-HIS-Part II
Record Dates: First submitted 2020-05-15; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2019-06

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus | interventions — Histamine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Single-blind, single-group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Histamine and placebo skin pricks (Other): Each subject will receive the same histamine (10 mg/ml) and control (saline) skin prick on the right and left forearm on both study visits, to allow an intra-individual comparison
  Interventions: Procedure: Histamine 10 mg/ml skin prick; Procedure: Placebo (saline) skin prick

INTERVENTIONS:
Procedure: Histamine 10 mg/ml skin prick — Skin prick through 5 µL histamine diHCl (10 mg/ml)
Procedure: Placebo (saline) skin prick — Skin prick through 5 µL saline (0.9% NaCl)

SUMMARY:
To evaluate the inter-arm and inter-period reproducibility of the dermal blood flow response induced by a skin prick of histamine, subjects will receive histamine (10 mg/ml) and negative control skin pricks on the volar surface of both forearms during two subsequent study visits to allow an intra-individual comparison. Changes in dermal blood flow will be measured during the hour after the skin pricks with laser Doppler and/or laser speckle contrast imaging.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a white male ≥ 18 and ≤ 45 years of age at the time of screening
* Subject is a nonsmoker for at least 6 months prior to the study start
* Subject has a body mass index ≥ 18 and ≤ 30 kg/m2
* Subject has a clear increase in histamine-induced dermal blood flow
* Subject is judged to be in good health on the basis of medical history, physical examination and vital signs
* Subject understands the procedures and agrees to comply with them for the entire length of the study by giving written informed consent

Exclusion Criteria:

* Subject has excessive hair growth on the volar surface of the forearm
* Subject has a past or present history of diffuse dermatological conditions including eczema, scleroderma, psoriasis, urticaria, dermatographism and dermatitis
* Subject has any abnormality on the skin of the forearm, possibly interfering with the study assessments including tattoos, keloids, tumors, ulcers, burns, flaps and grafts
* Subject cannot avoid excessive tanning (any exposure to sunlight or a tanning bed which would cause a sunburn reaction) throughout the study and cannot cover the forearms 24 hours before and after each study visit
* Subject currently uses lotions, oils, depilatory preparations, makeup or other topical treatments on the arms and on a regular basis which cannot be discontinued for the duration of the study; subject has used any topical treatments within 7 days of the start of the study
* Subject has a past or present history of (symptomatic) asthma
* Subject has a history of severe allergic reactions to food or drugs or adverse experiences of a serious nature related to the administration of either a marketed or investigational drug, including histamine
* Subject currently uses any prescription or nonprescription drugs on a regular basis which cannot be discontinued for the duration of the study; subject has used any prescription or nonprescription medication within 14 days of the start of the study
* Subject is a habitual and heavy consumer of coffee or caffeinated beverages (more than approximately 4 cups of tea, coffee or cola per day) at the time of the study. Subjects who have reduced their consumption to ≤ 4 cups per day at least 1 week prior to enrollment may participate. Subjects who cannot refrain from caffeinated beverages 24 hours before the study visit;
* Subject is unable to refrain from drinking alcohol 24 hours prior to histamine application, is currently a regular user (including "recreational use") of any illicit drugs, or has a history of drug (including alcohol) abuse. A drug screen will include amphetamines/ methamphetamines, methylenedioxymethamphetamine, benzodiazepines, barbiturates, cocaine, cannabis, tricyclic antidepressants, methadone and opiates
* Subject cannot refrain from being around second hand smoke 24 hours prior to histamine application or uses nicotine-containing products. Ex-smokers should have ceased smoking at least 6 months prior to screening
* Subject has any of the following vital sign measurements at screening: heart rate ≤ 40 or ≥ 100 beats/min, diastolic blood pressure ≤ 50 or ≥ 89 mmHg and/or systolic Blood Pressure ≤ 90 or ≥ 139 mmHg
* Subject has been involved in testing an investigational drug in another clinical study within the last 4 weeks or 5 half-lives
* Subject has evidence of a clinically significant active infection, fever of 38°C or above at the time of the study visits
* Subject has a history or current cardiovascular, respiratory, hepatic, renal, gastrointestinal or neurological disorders capable of significantly altering the absorption, metabolism or elimination of drugs
* Subject is in a situation or has a condition, which, in the opinion of the investigator, may interfere with safe and optimal participation in the study
* Subject has a history of any illness or disorder, which, in the opinion of the investigator, might confound the results of the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Change in dermal blood flow induced by histamine skin pricks, compared to baseline and placebo in terms of inter-period and inter-arm reproducability | The dermal blood flow will be assessed before (baseline) and every 5 minutes during the hour following the skin pricks

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Pharmacology, Leuven, Belgium